CLINICAL TRIAL: NCT07225673
Title: Feasibility and Effectiveness of Therapy Together: An Intensive Upper Limb Therapy Program for Young Children With Cerebral Palsy and Their Caregivers
Brief Title: Feasibility and Effectiveness of Therapy Together
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Scottish Rite Hospital for Children (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-1211
Record Dates: First submitted 2025-11-04; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 4 hour group (Active Comparator): The 4-hour group completed 32 hours in clinic and 24 hours at home (30 minutes per day) to complete the Therapy Together program.
  Interventions: Behavioral: Therapy Together - 4 hour group
- 1 hour group (Active Comparator): The 1-hour group completed 8 hours of in-clinic therapy and 48 hours of home-based activities (1 hour per day) to complete the Therapy Together program.
  Interventions: Behavioral: Therapy Together - 1 hour group

INTERVENTIONS:
Behavioral: Therapy Together - 4 hour group — a caregiver partnered constraint induced movement therapy program
  Arms: 4 hour group
Behavioral: Therapy Together - 1 hour group — a caregiver partnered constraint induced movement therapy program
  Arms: 1 hour group

SUMMARY:
this study proposes to compare the feasibility and effectiveness of 2 methods of delivery of Therapy Together, a caregiver and child intensive upper limb therapy program for children with CP and children at risk for developing CP ages 3 months - 4 years 11 months.

DETAILED DESCRIPTION:
One group will complete 32 hours onsite (4 hour weekly sessions) and 30 minutes of therapeutic activity at home, and the second group will complete 8 hours onsite and 1 hour of therapeutic activity at home. Both groups will aim to complete 56 hours of the intervention.

The Therapy Together program includes caregiver education and coaching on implementing therapeutic activities that are play-based, age-appropriate, and tailored to meet goals to improve arm/hand function. The child and caregiver complete 8 coaching sessions. The first 7 intervention visits focus on constraint-induced movement therapy (CIMT) and the final intervention visit focuses on bimanual therapy (use of two hands).

ELIGIBILITY:
Inclusion Criteria:

* present with asymmetric hand
* at risk for developing CP or children that have been diagnosed with CP
* must be able to visually attend to objects
* demonstrate an interest in objects
* attempt to reach for or grasp them with the impaired upper extremity

Exclusion Criteria:

* uncontrolled epilepsy
* significant visual impairment
* severe behavioral problems
* inability to complete the assessment protocol

Ages: 3 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Estimated)
Dates: Start 2020-01-02 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mini-Assisting Hand Assessment | pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention]
  The Mini-Assisting Hand Assessment is an observation-based, criterion-referenced assessment that assesses bimanual hand function for children with cerebral palsy aged 8-18 months (measured in logits/units)
Assisting Hand Assessment | pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Assisting Hand Assessment is an observation-based, criterion-referenced assessment that assess bimanual hand function for children with cerebral palsy, aged 18 months-12 years (measured in logits/units)

SECONDARY OUTCOMES:
Canadian Occupational Performance Measure | pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Canadian Occupational Performance Measure is an interview-based assessment of self-perception of performance of everyday living activities (measured on a scale from 1-10)
Developmental Assessment for Young Children, Second Edition (DAYC-2) | pre-intervention (within 2 weeks of start of intervention), and within 2 weeks of post-intervention
  The Developmental Assessment for Young Children is an interview and observation based norm-referenced developmental assessment (raw scores 0 or 1, converted to standard scores)
Weekly Caregiver Log | weekly for 8 weeks
  The caregiver log includes feasibility (time), stress, and impact on unilateral and bimanual hand function measured using a likert scale of 1-4

CONTACTS AND LOCATIONS:
Overall Officials: Angela Shierk, Principal Investigator — Scottish Rite for Children
Locations (1):
- Scottish Rite for Children, Frisco, Texas, United States

IPD SHARING:
Plan to Share IPD: No